CLINICAL TRIAL: NCT02682056
Title: Glucose Measurement Using Microneedle Patches
Acronym: GUMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Eric Felner, MD, MSCR, MD, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00075816
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Diabetes
Keywords: Pediatrics; Endocrinology; Adolescent; Microneedle
MeSH Terms: conditions — Diabetes Mellitus | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Study Arm (Other): Children and adolescents with diabetes will have blood glucose levels tested using microneedle patches, intravenous (IV) catheter draw, and lancet.
  Interventions: Device: Microneedle patch; Device: Intravenous (IV) catheter; Device: Lancet

INTERVENTIONS:
Device: Microneedle patch — The microneedle patch will collect interstitial fluid to be tested for glucose level. The microneedles are made from biocompatible polymers or metal. Participants will have fasting glucose levels measured four times, on an hourly basis, during the study visit.
Device: Intravenous (IV) catheter — The intravenous (IV) catheter will collect venous blood to be tested for glucose level. Participants will have fasting glucose levels measured four times, on an hourly basis, during the study visit.
Device: Lancet — The lancet will collect capillary blood to be tested for glucose level. Participants will have fasting glucose levels measured four times, on an hourly basis, during the study visit.

SUMMARY:
This study will compare three glucose measurement techniques among diabetic children and adolescents. The study seeks to determine if a microneedle patch (made from biocompatible polymers or metal), versus a lancet or intravenous catheter, would be a preferable option for monitoring glucose levels among the diabetic pediatric population.

DETAILED DESCRIPTION:
Fifteen children and adolescents with diabetes will be tested for their glucose measurements comparing interstitial fluid collected via a microneedle patch (made from biocompatible polymers or metal), versus the standard of care blood sample (lancet), and lab grade blood draw (intravenous catheter). Samples will be taken hourly from all three devices for four hours. All four measurements will be compared against each other to see how close they are with measuring the glucose values. Each participant will be asked to rate their apprehension prior to receiving each method for blood or interstitial fluid collection as well as the pain associated with each method immediately after collection.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes diagnosis

Exclusion Criteria:

* no exclusion criteria are specified

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Felner, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between December 2017 and January 2018 from the Emory Children's Center and Children's Healthcare of Atlanta, in Atlanta, Georgia.
Groups:
- Children Having Glucose Levels Tested Through Three Methods: Children and adolescents with diabetes having blood glucose levels tested using microneedle patches, intravenous (IV) catheter draw, and lancet. Sample collection with the different methods will occur simultaneously four times, on an hourly basis, during a single study visit.
Period: Overall Study
Arm/Group | Children Having Glucose Levels Tested Through Three Methods
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Children Having Glucose Levels Tested Through Three Methods: Children and adolescents with diabetes having blood glucose levels tested using microneedle patches, intravenous (IV) catheter draw, and lancet.
Arm/Group | Children Having Glucose Levels Tested Through Three Methods
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Glucose Level
Description: Participants had their glucose levels tested through three different methods. Interstitial glucose levels was assessed using a microneedles patch. Blood glucose levels were collected via the lancet and intravenous (IV) collection methods.
Time Frame: Baseline (Hour 1), Hour 2, Hour 3, Hour 4
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Microneedle: Microneedle patches were used to collect interstitial fluid for glucose testing. Participants had fasting glucose levels measured four time, on an hourly basis, during the study visit.
- Lancet: Lancets were used to collect capillary blood for glucose testing. Participants had fasting glucose levels measured four time, on an hourly basis, during the study visit.
- Intravenous Catheter: Intravenous catheters were used to collect venous blood for glucose testing. Participants had fasting glucose levels measured four time, on an hourly basis, during the study visit.
Arm/Group | Microneedle | Lancet | Intravenous Catheter
Number analyzed (Participants) | 15 | 15 | 15
mg/dL
  Baseline/Hour 1 | 137 (119) | 174.5 (58) | 160.9 (58)
  Hour 2 | 155 (78) | 271.4 (91) | 227.3 (65)
  Hour 3 | 256 (224) | 270.4 (82) | 270.4 (82)
  Hour 4 | 285 (126) | 276.4 (122.9) | 251.5 (122.9)

2. Secondary Outcome: Apprehension Level Assessed by Apprehension Visual Analog Scale (VAS)
Description: Participants completed a Visual Analog Scale (VAS) to report the level of apprehension they felt regarding each method of sample collection. Participants will mark on a line scale (between not afraid and very afraid) to indicate fear level when a sample is collected. The range is from 0-100 mm with 0 mm indicating no apprehension and 100 mm indicating the most apprehension.
Time Frame: Baseline ( Hour 1), Hour 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microneedle | Lancet | Intravenous Catheter
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline/Hour 1 | 24.1 (23.0) | 5.8 (16.9) | 30.8 (24.7)
  Hour 4 | 12.2 (14.1) | 4.9 (15.3) | 24.4 (20.6)

3. Secondary Outcome: Pain Level Assessed by Pain Visual Analog Scale (VAS)
Description: Participants completed a Visual Analog Scale (VAS) to report the level of pain they felt regarding each method of sample collection. Participants marked on a line scale (between no pain and worst pain ever) to indicate pain level when a sample is collected. The range is from 0-100 mm with 0 mm indicating no pain and 100 mm indicating the most extreme pain.
Time Frame: Baseline ( Hour 1), Hour 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Microneedle | Lancet | Intravenous Catheter
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline/Hour 1 | 22.5 (22.0) | 5.8 (16.9) | 33.4 (24.3)
  Hour 4 | 11.2 (13.5) | 4.4 (14.4) | 26.8 (21.1)

ADVERSE EVENTS:
Time Frame: Information about adverse events were collected from the time the study assessments began (Hour 1 on study Day 1) through the end of study procedures on study Day 1.
Arm/Group | Microneedle | Lancet | Intravenous Catheter
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT02682056/Prot_SAP_000.pdf